CLINICAL TRIAL: NCT04534972
Title: Strategy to Avoid Excessive Oxygen in Major Burn Patients (SAVE-O2)
Brief Title: Strategy to Avoid Excessive Oxygen in Major Burn Patients
Acronym: SAVE-O2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-2799
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Wounds and Injury; Disease Attributes; Pathologic Processes
Keywords: hypoxia; hyperoxia; burn; critical illness; supplemental oxygen; oxygenation; SpO2; PaO2; FiO2; normoxia; hypoxemia; hyperoxemia; normoxemia
MeSH Terms: conditions — Critical Illness; Wounds and Injuries; Disease Attributes; Pathologic Processes; Hypoxia; Hyperoxia; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation (No Intervention): The control (pre-implementation) group will be burn patients admitted to the burn unit in ICU during the site's control period of the stepped-wedge implementation process (up to 22 months).
- Post-Implementation Targeting Normoxemia in Burn ICU (Active Comparator): The intervention (post-implementation) group will be patients admitted to the burn unit in ICU during the targeting normoxemia intervention period of the stepped-wedge design implementation process (up to 19 months).
  Interventions: Other: Targeting Normoxemia (SpO2 90-96%; PaO2 60-100 mmHg)

INTERVENTIONS:
Other: Targeting Normoxemia (SpO2 90-96%; PaO2 60-100 mmHg) — Post-implementation of targeted normoxemia through oxygen titration for individual patients. Intervention for treatment of hypoxemia will follow usual local practice. Interventions for treatment of hyperoxemia (SpO2 >96% or PaO2 > 100 mmHg) will involve down titration of FiO2 (or supplemental oxygen for non-mechanically ventilated patients) within a time frame based on local site preferences-typically in increments of no greater than 0.10 until goal oxygenation in the normoxemia range is achieved (including room air [no supplemental oxygen] for non-mechanically ventilated patients).
  Arms: Post-Implementation Targeting Normoxemia in Burn ICU

SUMMARY:
The objective is to determine the effectiveness of a multimodal educational intervention to reduce supplemental oxygen use in major burn patients. Investigators will also evaluate the safety and clinical effectiveness of the more targeted use of oxygen therapy.

DETAILED DESCRIPTION:
Oxygen therapy has undisputed importance in the care of critically ill patients to prevent secondary complications related to hypoxemia. Although routine, the practice of excessive over-oxygenation may be harmful. An expert panel was convened and developed the strong consensus to target normoxemia at an oxygen saturation (SpO2) range of 90-96%, an arterial oxygen (PaO2) range of 60-100 mmHg (when applicable), and a fraction of inspired oxygen (FiO2) of 21% for mechanically ventilated patients or room air for nonmechanically ventilated patients.

Specific Aim: The purpose of this study is to determine the effectiveness of a multimodal educational intervention to reduce supplemental oxygen use in major burn patients. Investigators will also evaluate the safety and clinical effectiveness of the more targeted use of oxygen therapy.

Hypotheses: Clinical efforts to through a multimodal educational intervention will:

1. Improve the proportion of time spent within target normoxemia thresholds (oxygen saturation [SpO2] 90-96% and/or arterial oxygen [PaO2] 60-100 mmHg [when applicable])
2. Limiting use of excessive supplemental oxygen
3. Reduce exposure to hyperoxemia without a substantive increase in hypoxemic episodes or adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute thermal burn injury who meet the criteria for entry into the state or national burn data repository
* Admission to burn unit within 24 hours of burn injury

Exclusion Criteria:

* Age <18 years
* Prisoners
* Known pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Supplemental Oxygen Free Days (SOFD) | up to 28 days
  Number of days alive and not on supplemental oxygen during the index hospitalization (0 days [worst outcome] to 28 days [best outcome])

SECONDARY OUTCOMES:
Hospital-Free Days to day 90 (HFD90) | up to 90 days
  Number of days alive and outside the hospital (0 days [worst outcome] to 90 days [best outcome])
In-hospital Mortality to day 90 | up to 90 days
  Dichotomous vital status (survived or died) at hospital discharge or day 90, whichever is first
Time to Mortality to day 90 | up to 90 days
  Vital status and date of death censored at hospital discharge or day 90, whichever is first
Ventilator Free Days (VFD) to day 28 | up to 28 days
  Ventilator Free days = Days off ventilator (0 VFD [worst outcome] to 28 VFD [best outcome])
Time to Room air | up to 90 days
  Duration of supplemental oxygen (FiO2 = 0.21 or room air)
Time to Burn Wound Healing | up to 90 days
  Wound closure of >90% of the original burn or time to grafting (for non-full thickness wounds)
Discharge Disposition | up to 90 days
  Defined as home (return to prior level of care) or facility (e.g., acute rehab, skilled nursing facility)
Amount of Supplemental Oxygen Administered | up to 90 days
  Total estimated oxygen volume while in the burn until after hospital arrival
Duration of Time on Normoxemia Protocol Target | up to 90 days
  Defined as SpO2 90-96% or receiving no supplemental oxygen (FiO2 0.21 or room air) while in the burn unit
Proportion of Participants Receiving High Levels of Supplemental Oxygen | up to 90 days
  FiO2>0.40 or >4 liters per minute for >2 hours while in the burn unit [excludes time in the operating room]
Duration of Time Receiving High Levels of Supplemental Oxygen | up to 90 days
  FiO2>0.40 or >4 liters per minute while in the burn unit
Duration of Time Receiving No Supplemental Oxygen | up to 90 days
  FiO2 0.21 or room air while in the burn unit
Incidence of Hypoxemic Event (SpO2<88%) | up to 90 days
  SpO2 saturation below 88% while in the burn unit
Duration of Hypoxemic Events (SpO2<88%) | up to 90 days
  SpO2 saturation below 88% while in the burn unit
Incidence of Hyperoxemic Event (SpO2>96%) | up to 90 days
  SpO2 saturation above 96% while in the burn unit
Duration of Hyperoxemic Event (SpO2>96%) | up to 90 days
  SpO2 saturation above 96% while in the burn unit

CONTACTS AND LOCATIONS:
Overall Officials: Adit Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Alabama-Birmingham Medical Center, Birmingham, Alabama
  - University of Colorado, Aurora, Colorado
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Army Institute of Surgical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leverve XM. To cope with oxygen: a long and still tumultuous story for life. Crit Care Med. 2008 Feb;36(2):637-8. doi: 10.1097/CCM.0B013E31816296AD. No abstract available. PMID 18216624
- [Background] Damiani E, Adrario E, Girardis M, Romano R, Pelaia P, Singer M, Donati A. Arterial hyperoxia and mortality in critically ill patients: a systematic review and meta-analysis. Crit Care. 2014 Dec 23;18(6):711. doi: 10.1186/s13054-014-0711-x. PMID 25532567
- [Background] Panwar R, Capellier G, Schmutz N, Davies A, Cooper DJ, Bailey M, Baguley D, Pilcher V, Bellomo R. Current oxygenation practice in ventilated patients-an observational cohort study. Anaesth Intensive Care. 2013 Jul;41(4):505-14. doi: 10.1177/0310057X1304100412. PMID 23808511
- [Background] Suzuki S, Eastwood GM, Peck L, Glassford NJ, Bellomo R. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care. 2013 Oct;28(5):647-54. doi: 10.1016/j.jcrc.2013.03.010. Epub 2013 May 15. PMID 23683560
- [Background] Rachmale S, Li G, Wilson G, Malinchoc M, Gajic O. Practice of excessive F(IO(2)) and effect on pulmonary outcomes in mechanically ventilated patients with acute lung injury. Respir Care. 2012 Nov;57(11):1887-93. doi: 10.4187/respcare.01696. Epub 2012 May 15. PMID 22613692
- [Background] Parke RL, Eastwood GM, McGuinness SP; George Institute for Global Health; Australian and New Zealand Intensive Care Society Clinical Trials Group. Oxygen therapy in non-intubated adult intensive care patients: a point prevalence study. Crit Care Resusc. 2013 Dec;15(4):287-93. PMID 24289510
- [Background] Iscoe S, Beasley R, Fisher JA. Supplementary oxygen for nonhypoxemic patients: O2 much of a good thing? Crit Care. 2011;15(3):305. doi: 10.1186/cc10229. Epub 2011 Jun 30. PMID 21722334
- [Background] Panwar R, Young P, Capellier G. Conservative oxygen therapy in mechanically ventilated patients. Crit Care Med. 2014 Sep;42(9):e630-1. doi: 10.1097/CCM.0000000000000439. No abstract available. PMID 25126814
- [Background] de Graaff AE, Dongelmans DA, Binnekade JM, de Jonge E. Clinicians' response to hyperoxia in ventilated patients in a Dutch ICU depends on the level of FiO2. Intensive Care Med. 2011 Jan;37(1):46-51. doi: 10.1007/s00134-010-2025-z. Epub 2010 Sep 28. PMID 20878146
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Pannu SR. Too Much Oxygen: Hyperoxia and Oxygen Management in Mechanically Ventilated Patients. Semin Respir Crit Care Med. 2016 Feb;37(1):16-22. doi: 10.1055/s-0035-1570359. Epub 2016 Jan 28. PMID 26820270
- [Background] Kallet RH, Branson RD. Should Oxygen Therapy Be Tightly Regulated to Minimize Hyperoxia in Critically Ill Patients? Respir Care. 2016 Jun;61(6):801-17. doi: 10.4187/respcare.04933. PMID 27235315
- [Background] Hafner S, Beloncle F, Koch A, Radermacher P, Asfar P. Hyperoxia in intensive care, emergency, and peri-operative medicine: Dr. Jekyll or Mr. Hyde? A 2015 update. Ann Intensive Care. 2015 Dec;5(1):42. doi: 10.1186/s13613-015-0084-6. Epub 2015 Nov 19. PMID 26585328
- [Background] Singh V, Devgan L, Bhat S, Milner SM. The pathogenesis of burn wound conversion. Ann Plast Surg. 2007 Jul;59(1):109-15. doi: 10.1097/01.sap.0000252065.90759.e6. PMID 17589272
- [Background] Cancio LC, Barillo DJ, Kearns RD, Holmes JH 4th, Conlon KM, Matherly AF, Cairns BA, Hickerson WL, Palmieri T. Guidelines for Burn Care Under Austere Conditions: Surgical and Nonsurgical Wound Management. J Burn Care Res. 2017 Jul/Aug;38(4):203-214. doi: 10.1097/BCR.0000000000000368. No abstract available. PMID 27355660
- [Background] Palmieri TL, Przkora R, Meyer WJ 3rd, Carrougher GJ. Measuring burn injury outcomes. Surg Clin North Am. 2014 Aug;94(4):909-16. doi: 10.1016/j.suc.2014.05.010. PMID 25085096
- [Background] Kao Y, Loh EW, Hsu CC, Lin HJ, Huang CC, Chou YY, Lien CC, Tam KW. Fluid Resuscitation in Patients With Severe Burns: A Meta-analysis of Randomized Controlled Trials. Acad Emerg Med. 2018 Mar;25(3):320-329. doi: 10.1111/acem.13333. Epub 2017 Nov 11. PMID 29024269
- [Background] Helmerhorst HJ, Roos-Blom MJ, van Westerloo DJ, de Jonge E. Association Between Arterial Hyperoxia and Outcome in Subsets of Critical Illness: A Systematic Review, Meta-Analysis, and Meta-Regression of Cohort Studies. Crit Care Med. 2015 Jul;43(7):1508-19. doi: 10.1097/CCM.0000000000000998. PMID 25855899
- [Background] Austin MA, Wills KE, Blizzard L, Walters EH, Wood-Baker R. Effect of high flow oxygen on mortality in chronic obstructive pulmonary disease patients in prehospital setting: randomised controlled trial. BMJ. 2010 Oct 18;341:c5462. doi: 10.1136/bmj.c5462. PMID 20959284
- [Background] Chi JH, Knudson MM, Vassar MJ, McCarthy MC, Shapiro MB, Mallet S, Holcroft JJ, Moncrief H, Noble J, Wisner D, Kaups KL, Bennick LD, Manley GT. Prehospital hypoxia affects outcome in patients with traumatic brain injury: a prospective multicenter study. J Trauma. 2006 Nov;61(5):1134-41. doi: 10.1097/01.ta.0000196644.64653.d8. PMID 17099519
- [Background] Panwar R, Hardie M, Bellomo R, Barrot L, Eastwood GM, Young PJ, Capellier G, Harrigan PW, Bailey M; CLOSE Study Investigators; ANZICS Clinical Trials Group. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Jan 1;193(1):43-51. doi: 10.1164/rccm.201505-1019OC. PMID 26334785
- [Background] ICU-ROX Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Mackle D, Bellomo R, Bailey M, Beasley R, Deane A, Eastwood G, Finfer S, Freebairn R, King V, Linke N, Litton E, McArthur C, McGuinness S, Panwar R, Young P; ICU-ROX Investigators the Australian and New Zealand Intensive Care Society Clinical Trials Group. Conservative Oxygen Therapy during Mechanical Ventilation in the ICU. N Engl J Med. 2020 Mar 12;382(11):989-998. doi: 10.1056/NEJMoa1903297. Epub 2019 Oct 14. PMID 31613432
- [Background] Schmidt B, Whyte RK, Asztalos EV, Moddemann D, Poets C, Rabi Y, Solimano A, Roberts RS; Canadian Oxygen Trial (COT) Group. Effects of targeting higher vs lower arterial oxygen saturations on death or disability in extremely preterm infants: a randomized clinical trial. JAMA. 2013 May 22;309(20):2111-20. doi: 10.1001/jama.2013.5555. PMID 23644995
- [Background] Stockinger ZT, Mcswain NE Jr. Prehospital supplemental oxygen in trauma patients: its efficacy and implications for military medical care. Mil Med. 2004 Aug;169(8):609-12. doi: 10.7205/milmed.169.8.609. PMID 15379072
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023
- [Background] Stub D, Smith K, Bernard S, Nehme Z, Stephenson M, Bray JE, Cameron P, Barger B, Ellims AH, Taylor AJ, Meredith IT, Kaye DM; AVOID Investigators. Air Versus Oxygen in ST-Segment-Elevation Myocardial Infarction. Circulation. 2015 Jun 16;131(24):2143-50. doi: 10.1161/CIRCULATIONAHA.114.014494. Epub 2015 May 22. PMID 26002889
- [Background] Suzuki S, Eastwood GM, Glassford NJ, Peck L, Young H, Garcia-Alvarez M, Schneider AG, Bellomo R. Conservative oxygen therapy in mechanically ventilated patients: a pilot before-and-after trial. Crit Care Med. 2014 Jun;42(6):1414-22. doi: 10.1097/CCM.0000000000000219. PMID 24561566
- [Background] Eastwood GM, Peck L, Young H, Suzuki S, Garcia M, Bellomo R. Intensive care clinicians' opinion of conservative oxygen therapy (SpO(2) 90-92%) for mechanically ventilated patients. Aust Crit Care. 2014 Aug;27(3):120-5. doi: 10.1016/j.aucc.2013.11.004. Epub 2013 Dec 24. PMID 24369915
- [Background] Helmerhorst HJ, Schultz MJ, van der Voort PH, Bosman RJ, Juffermans NP, de Jonge E, van Westerloo DJ. Self-reported attitudes versus actual practice of oxygen therapy by ICU physicians and nurses. Ann Intensive Care. 2014 Jul 25;4:23. doi: 10.1186/s13613-014-0023-y. eCollection 2014. PMID 25512878
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Baker DW, Persell SD. Criteria for waiver of informed consent for quality improvement research. JAMA Intern Med. 2015 Jan;175(1):142-3. doi: 10.1001/jamainternmed.2014.6977. No abstract available. PMID 25560946
- [Background] McKinney RE Jr, Beskow LM, Ford DE, Lantos JD, McCall J, Patrick-Lake B, Pletcher MJ, Rath B, Schmidt H, Weinfurt K. Use of altered informed consent in pragmatic clinical research. Clin Trials. 2015 Oct;12(5):494-502. doi: 10.1177/1740774515597688. Epub 2015 Sep 15. PMID 26374677
- [Background] Douin DJ, Schauer SG, Anderson EL, Jones J, DeSanto K, Cunningham CW, Bebarta VS, Ginde AA. Systematic review of oxygenation and clinical outcomes to inform oxygen targets in critically ill trauma patients. J Trauma Acute Care Surg. 2019 Oct;87(4):961-977. doi: 10.1097/TA.0000000000002392. PMID 31162333
- [Background] BOOST II United Kingdom Collaborative Group; BOOST II Australia Collaborative Group; BOOST II New Zealand Collaborative Group; Stenson BJ, Tarnow-Mordi WO, Darlow BA, Simes J, Juszczak E, Askie L, Battin M, Bowler U, Broadbent R, Cairns P, Davis PG, Deshpande S, Donoghoe M, Doyle L, Fleck BW, Ghadge A, Hague W, Halliday HL, Hewson M, King A, Kirby A, Marlow N, Meyer M, Morley C, Simmer K, Tin W, Wardle SP, Brocklehurst P. Oxygen saturation and outcomes in preterm infants. N Engl J Med. 2013 May 30;368(22):2094-104. doi: 10.1056/NEJMoa1302298. Epub 2013 May 5. PMID 23642047
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Derived] Douin DJ, Rice JD, Xiao M, Jackson CL, Anderson EL, Cheng AC, Cwik J, Beaty LE, Wild JL, Beyene RT, Britton GW, Corcos AC, Dale EL, Hwang J, Jansen JO, Self WH, Slater JC, Steinwand A, Wiktor AJ, Ziembicki J, Schauer SG, Bebarta VS, Cancio L, Ginde AA; Strategy to Avoid Excessive Oxygen (SAVE-O2) Investigators. Effect of targeting normoxemia on supplemental oxygen-free days for adults with acute thermal burns: A stepped wedge cluster randomized clinical trial. J Trauma Acute Care Surg. 2025 Oct 1;99(4):619-627. doi: 10.1097/TA.0000000000004712. Epub 2025 Jul 3. PMID 40604863